CLINICAL TRIAL: NCT00508027
Title: Phase I/II Study of Simvastatin (Zocor) Therapy in Sickle Cell Disease
Brief Title: Simvastatin (Zocor) Therapy in Sickle Cell Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Carolyn Hoppe, Associate Hematologist, UCSF Benioff Children's Hospital Oakland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01FD003080-01A1 (FDA)
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Results first posted 2013-08-16 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-08

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; simvastatin; statin drugs; nitric oxide donors; vascular injury
MeSH Terms: conditions — Anemia, Sickle Cell; Vascular System Injuries | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Simvastatin, Dose Escalation (Other): There are no arms in this study. Simvastatin will be given in a dose-escalating fashion to 3 sequential dosage groups (20 mg/day, 40 mg/day, 80 mg/day).
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Comparison of 3 dosages of simvastatin given in a dose-escalating fashion. 20 mg, 40 mg, or 80 mg PO QD x 21 days followed by a drug taper x 4 days.
  Other Names: Zocor

SUMMARY:
Recent clinical and experimental data indicate that statins have effects beyond cholesterol lowering that may be beneficial in sickle cell disease by protecting the vascular endothelium. Statins have been shown to attenuate endothelial dysfunction through their anti-inflammatory, anti-oxidant and anti-thrombotic properties. This phase I/II dose-escalating trial is designed to assess the safety and potential clinical efficacy of oral simvastatin (Zocor)in adolescents and adults with sickle cell disease (SCD).

DETAILED DESCRIPTION:
Although statins have been used extensively for their cholesterol-lowering effects, recent clinical and experimental data indicate that statins regulate yet other processes, many of which play a major role in sickle cell disease (SCD). Independent of their cholesterol-lowering effects, statins have been shown to prevent damage to blood vessels in several ways, through upregulation of endothelial nitric oxide (NO)and decreased inflammation. Numerous studies documenting the protective effects of statins, together with data showing the therapeutic role of NO in SCD, provide the basis for investigating the potential clinical benefit of simvastatin in SCD.

Data supporting the safety and tolerability of simvastatin in patients with SCD are now needed. For this phase I/II dose-escalation study of oral simvastatin in SCD, we propose the following specific aims:

1. To obtain preliminary efficacy data on the effects of oral simvastatin on plasma biomarkers of endothelial injury in patients with SCD, and
2. To assess the safety and tolerability of oral simvastatin in patients with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of sickle cell disease (HbSS, SC or Sβ-thalassemia)
* Age greater than or equal to thirteen years
* Weight greater than or equal to 35 kg

Exclusion Criteria:

* Renal dysfunction (Serum Creatinine > 1.5 UNL)
* Hepatic dysfunction (ALT > 2X UNL)
* Pretreatment total cholesterol < 100 mg/dL or triglycerides < 30 mg/dL
* Pretreatment baseline creatine kinase >1X UNL (215 U/L)
* Pregnancy/lactation
* RBC transfusion in the last 30 days
* Vaso-Occlusive Event needing hospitalization in the past 30 days
* Treatment with any statin drugs within the past 30 days
* Treatment with drugs having known metabolic interactions with statin drugs (e.g. cytochrome P450 3A4 metabolism), including ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, azithromycin, niacin (nicotinic acid), digoxin, coumadin, sildenafil or amiodarone within the past 30 days
* Treatment (past or present) with amiodarone
* Musculoskeletal disorder associated with an elevated creatine kinase level
* Past or present history of substance abuse (alcohol, cocaine, amphetamines, heroin, PCP)
* Allergy to statins

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn C Hoppe, M.D., Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Children's Hospital and Research Center Oakland, Oakland, California, United States

REFERENCES:
- [Background] Hebbel RP. Extracorpuscular factors in the pathogenesis of sickle cell disease. Am J Pediatr Hematol Oncol. 1982 Fall;4(3):316-9. PMID 7149170
- [Background] Hebbel RP. Perspectives series: cell adhesion in vascular biology. Adhesive interactions of sickle erythrocytes with endothelium. J Clin Invest. 1997 Jun 1;99(11):2561-4. doi: 10.1172/JCI119442. No abstract available. PMID 9169483
- [Background] Hebbel RP. Special issue of Microcirculation: examination of the vascular pathobiology of sickle cell anemia. Foreword. Microcirculation. 2004 Mar;11(2):99-100. No abstract available. PMID 15280085
- [Background] Kaul DK, Liu XD, Choong S, Belcher JD, Vercellotti GM, Hebbel RP. Anti-inflammatory therapy ameliorates leukocyte adhesion and microvascular flow abnormalities in transgenic sickle mice. Am J Physiol Heart Circ Physiol. 2004 Jul;287(1):H293-301. doi: 10.1152/ajpheart.01150.2003. Epub 2004 Mar 4. PMID 15001449
- [Background] Wood KC, Hebbel RP, Granger DN. Endothelial cell P-selectin mediates a proinflammatory and prothrombogenic phenotype in cerebral venules of sickle cell transgenic mice. Am J Physiol Heart Circ Physiol. 2004 May;286(5):H1608-14. doi: 10.1152/ajpheart.01056.2003. Epub 2004 Jan 2. PMID 14704223
- [Background] Belcher JD, Marker PH, Weber JP, Hebbel RP, Vercellotti GM. Activated monocytes in sickle cell disease: potential role in the activation of vascular endothelium and vaso-occlusion. Blood. 2000 Oct 1;96(7):2451-9. PMID 11001897
- [Background] Haffner SM, Alexander CM, Cook TJ, Boccuzzi SJ, Musliner TA, Pedersen TR, Kjekshus J, Pyorala K. Reduced coronary events in simvastatin-treated patients with coronary heart disease and diabetes or impaired fasting glucose levels: subgroup analyses in the Scandinavian Simvastatin Survival Study. Arch Intern Med. 1999 Dec 13-27;159(22):2661-7. doi: 10.1001/archinte.159.22.2661. PMID 10597756
- [Background] Laufs U, Wassmann S, Hilgers S, Ribaudo N, Bohm M, Nickenig G. Rapid effects on vascular function after initiation and withdrawal of atorvastatin in healthy, normocholesterolemic men. Am J Cardiol. 2001 Dec 1;88(11):1306-7. doi: 10.1016/s0002-9149(01)02095-1. No abstract available. PMID 11728362
- [Background] Hebbel RP, Vercellotti GM. The endothelial biology of sickle cell disease. J Lab Clin Med. 1997 Mar;129(3):288-93. doi: 10.1016/s0022-2143(97)90176-1. No abstract available. PMID 9042813
- [Background] Solovey A, Lin Y, Browne P, Choong S, Wayner E, Hebbel RP. Circulating activated endothelial cells in sickle cell anemia. N Engl J Med. 1997 Nov 27;337(22):1584-90. doi: 10.1056/NEJM199711273372203. PMID 9371854
- [Background] Solovey A, Gui L, Key NS, Hebbel RP. Tissue factor expression by endothelial cells in sickle cell anemia. J Clin Invest. 1998 May 1;101(9):1899-904. doi: 10.1172/JCI1932. PMID 9576754
- [Background] Reiter CD, Gladwin MT. An emerging role for nitric oxide in sickle cell disease vascular homeostasis and therapy. Curr Opin Hematol. 2003 Mar;10(2):99-107. doi: 10.1097/00062752-200303000-00001. PMID 12579034
- [Background] Gladwin MT, Crawford JH, Patel RP. The biochemistry of nitric oxide, nitrite, and hemoglobin: role in blood flow regulation. Free Radic Biol Med. 2004 Mar 15;36(6):707-17. doi: 10.1016/j.freeradbiomed.2003.11.032. PMID 14990351
- [Background] Platt OS. Sickle cell anemia as an inflammatory disease. J Clin Invest. 2000 Aug;106(3):337-8. doi: 10.1172/JCI10726. No abstract available. PMID 10930436
- [Background] Brown MD, Wick TM, Eckman JR. Activation of vascular endothelial cell adhesion molecule expression by sickle blood cells. Pediatr Pathol Mol Med. 2001 Jan-Feb;20(1):47-72. PMID 12673844
- [Background] Takemoto M, Liao JK. Pleiotropic effects of 3-hydroxy-3-methylglutaryl coenzyme a reductase inhibitors. Arterioscler Thromb Vasc Biol. 2001 Nov;21(11):1712-9. doi: 10.1161/hq1101.098486. PMID 11701455
- [Background] Corsini A, Bellosta S, Baetta R, Fumagalli R, Paoletti R, Bernini F. New insights into the pharmacodynamic and pharmacokinetic properties of statins. Pharmacol Ther. 1999 Dec;84(3):413-28. doi: 10.1016/s0163-7258(99)00045-5. PMID 10665838
- [Result] Hoppe C, Kuypers F, Larkin S, Hagar W, Vichinsky E, Styles L. A pilot study of the short-term use of simvastatin in sickle cell disease: effects on markers of vascular dysfunction. Br J Haematol. 2011 Jun;153(5):655-63. doi: 10.1111/j.1365-2141.2010.08480.x. Epub 2011 Apr 8. PMID 21477202
- See also: Children's Hospital and Research Center Oakland Official Website — http://www.childrenshospitaloakland.org
- See also: NHLBI Website - Sickle Cell Disease — http://www.nhlbi.nih.gov/health/dci/Diseases/Sca/SCA_WhatIs.html
- See also: Medline Plus: Sickle Cell Anemia — http://www.nlm.nih.gov/medlineplus/ency/article/000527.htm
- See also: CHO Library: Sickle Cell Disease Information — http://www.childrenshospitaloakland.org/healthcare/health_library.asp
- See also: CHO Sickle Cell Program: National Center for Sickle Cell Disease — http://www.childrenshospitaloakland.org/healthcare/depts/sickle_cell_center.asp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the study period (05/2006-09/2010), eligible adult and adolescent SCD subjects followed at the CHRCO Sickle Cell Center were approached about participation in this trial. Subjects were enrolled at "steady-state" (i.e., no acute illness or acute SCD-related complications) during a routine clinic visit.
Pre-assignment Details: There were no significant events following enrollment after inclusion and exclusion criteria were met.
Groups:
- Simvastatin, 3 Escalating Dose Groups: Simvastatin was given in a dose-escalating fashion to 3 sequential dose groups:
  dose level 1= 20 mg/day, dose level 2= 40 mg/day, dose level 3= 80 mg/day The number of subjects starting each dose level are new cohorts of subjects.
  Determination of clinical safety in the first dose level group was required in order to begin enrollment in the second dose level group and ultimately the third dose group. Enrollment in the third dose level was discontinued early due to newly reported FDA warnings regarding high dose (80mg/day) simvastatin.
Period: Dose Level 1
Arm/Group | Simvastatin, 3 Escalating Dose Groups
Started | 20 (The participants starting each dose period is a new cohort of subjects. 20 subjects started dose 1)
Completed | 12
Not Completed | 8
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2
Period: Dose Level 2
Arm/Group | Simvastatin, 3 Escalating Dose Groups
Started | 20 (The participants starting each dose period is a new cohort of subjects. 20 new subjects in dose 2)
Completed | 16
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Period: Dose Level 3
Arm/Group | Simvastatin, 3 Escalating Dose Groups
Started | 2 (enrollment discontinued due to FDA recommendations regarding high dose (80mg/day) simvastatin)
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 42 subjects started the study; of these,12 were withdrawn from the study and 30 completed the study: dose level 1 (n=16); dose level 2 (n=12), dose level 3 (n=2). Only those participants who completed the study were included in the final analyses (n=30).
Groups:
- Simvastatin, Dose Escalation: There are no arms in this study. Simvastatin will be given in a dose-escalating fashion to 3 sequential dosage groups (20 mg/day, 40 mg/day, 80 mg/day).
  Simvastatin : Comparison of 3 dosages of simvastatin given in a dose-escalating fashion.
  20 mg, 40 mg, or 80 mg PO QD x 21 days followed by a drug taper x 4 days.
Arm/Group | Simvastatin, Dose Escalation
Number analyzed (Participants) | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 25 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 30
Sickle cell genotype [Number; unit: participants]
  Homozygous Hb S (SS or S/beta0 thalassemia) | 20
  Compound heterozygous Hb S and Hb C (SC) | 10

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Change in Plasma NOx Levels
Description: Measurements of the levels of plasma nitric oxide metabolites (NOx), high sensitivity C-reactive protein (hs-CRP), interleukin-6 (IL-6), vascular cell adhesion molecule-1 (VCAM-1), tissue factor (TF) and vascular endothelial growth factor (VEGF)were performed before and after simvastatin treatment. Changes in mean plasma biomarker levels were assessed for each dose level; however, dose level 3 results were not analyzed, as only 2 subjects were enrolled in this dose group.
Time Frame: Baseline, 21 days
Population: All participants for whom plasma biomarker levels were recorded at baseline and 21 days
Measure: Mean (Standard Deviation); unit: micromolar
Groups:
- Simvastatin, Dose Level 1: All participants received 20mg simvastatin once daily
- Simvastatin, Dose Level 2: All participants received 40 mg of simvastatin once daily
- Simvastatin, Dose Level 3: subject received 80 mg daily; biomarker data were not collected for participants enrolled in Dose Level 3 (80mg/day) due to discontinuation for recent FDA restriction on daily dosage
Arm/Group | Simvastatin, Dose Level 1 | Simvastatin, Dose Level 2 | Simvastatin, Dose Level 3
Number analyzed (Participants) | 16 | 12 | 0
micromolar | 7 (1) | 19.7 (12) |
Statistical Analysis 1: Comparison: Simvastatin, Dose Level 1 vs Simvastatin, Dose Level 2; Ho: There is no change in plasma biomarker levels before and after simivastatin treatment. With 12 patients in each group and assuming a 5% risk of Type I error (two-tailed α = 0.05) and estimated SD for the change in NOx (or sVCAM-1) of 48%, power will be 80% to detect a 40% change from baseline for each group, and a 55% difference in the change in biomarker levels between dose groups. Matched paired t-tests were used to measure changes in biomarker levels from baseline; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 5.5, Standard Deviation 1.7

2. Other Pre Specified Outcome: Change in Plasma Hs-CRP Levels
Description: Change in plasma high sensitivity C-reactive protein levels in subjects treated with simvastatin
Time Frame: Baseline, 21 days
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Simvastatin, Dose Level 3: subject received 80 mg daily; only descriptive clinical data collected for participants enrolled in Dose Level 3 (80mg/day) due to discontinuation for recent FDA restriction on daily dosage
Arm/Group | Simvastatin, Dose Level 1 | Simvastatin, Dose Level 2 | Simvastatin, Dose Level 3
Number analyzed (Participants) | 16 | 12 | 0
mg/L | -7.7 (14.2) | -3.6 (4.8) |

3. Other Pre Specified Outcome: Change in Plasma IL-6 Levels
Description: Change in plasma IL-6 level after treatment with simvastatin
Time Frame: Baseline, 21 days
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Simvastatin, Dose Level 1 | Simvastatin, Dose Level 2 | Simvastatin, Dose Level 3
Number analyzed (Participants) | 16 | 12 | 0
pg/mL | -0.6 (0.9) | -0.3 (0.3) |

4. Other Pre Specified Outcome: Change in Plasma VEGF Levels
Description: Change in plasma vascular endothelial adhesion molecule-1 levels after treatment with simvastatin
Time Frame: Baseline, 21 days
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Dose Level 1: All participants received 20mg simvastatin once daily
- Dose Level 2: All participants received 40 mg of simvastatin once daily
Arm/Group | Dose Level 1 | Dose Level 2 | Simvastatin, Dose Level 3
Number analyzed (Participants) | 16 | 12 | 0
pg/mL | -164 (40) | -30 (20) |

5. Other Pre Specified Outcome: Change in Plasma VCAM1 Levels
Description: Change in plasma vascular cellular adhesion molecule-1 levels after treatment with simvastatin
Time Frame: Baseline, 21 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Simvastatin, Dose Level 1 | Simvastatin, Dose Level 2 | Simvastatin, Dose Level 3
Number analyzed (Participants) | 16 | 12 | 0
ng/mL | -44 (58) | -86 (103) |

6. Other Pre Specified Outcome: Change in Plasma TF Levels
Description: Change in plasma tissue factor (TF) levels after treatment with simvastatin
Time Frame: Baseline, 21 days
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Simvastatin, Dose Level 1 | Simvastatin, Dose Level 2 | Simvastatin, Dose Level 3
Number analyzed (Participants) | 16 | 12 | 0
pg/mL | -9 (32) | -36 (54) |

7. Primary Outcome: Change in Total Cholesterol Level
Description: Change in serum total cholesterol level after treatment with simvastatin
Time Frame: Baseline, 21 days
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Simvastatin, Dose Level 1: All participants received 20 mg of simvastatin once daily
- Simvastatin, Dose Level 3: Subjects received 80 mg daily. Data collected for only 2 participants enrolled in Dose Level 3 (80mg/day) due to discontinuation for recent FDA restriction on daily dosage"
Arm/Group | Simvastatin, Dose Level 1 | Simvastatin, Dose Level 2 | Simvastatin, Dose Level 3
Number analyzed (Participants) | 16 | 12 | 2
mg/dL | -16 (2) | -18 (10) | -18 (4)

8. Primary Outcome: Change in Hemoglobin Level
Description: Change in plasma hemoglobin (Hb) level after treatment with simvastatin
Time Frame: Baseline, 21 days
Measure: Mean (Standard Deviation); unit: gm/dL
Arm/Group | Simvastatin, Dose Level 1 | Simvastatin, Dose Level 2 | Simvastatin, Dose Level 3
Number analyzed (Participants) | 16 | 12 | 2
gm/dL | -0.2 (0.1) | 0.1 (0.2) | -0.4 (0.1)

9. Primary Outcome: Change in Serum Creatine Kinase Levels
Description: Change in serum creatine kinase (CK) levels after treatment with simvastatin
Time Frame: Baseline, 21 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Simvastatin, Dose Level 1 | Simvastatin, Dose Level 2 | Simvastatin, Dose Level 3
Number analyzed (Participants) | 16 | 12 | 2
U/L | 57 (88) | 20 (34) | 62 (20)

10. Primary Outcome: Change in Serum Alanine Transaminase (ALT) Levels
Description: Change in serum alanine transaminase (ALT) after treatment with simvastatin
Time Frame: Baseline, 21 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Simvastatin, Dose Level 1 | Simvastatin, Dose Level 2 | Simvastatin, Dose Level 3
Number analyzed (Participants) | 16 | 12 | 2
U/L | 4 (3) | 3 (4) | -3 (2)

11. Primary Outcome: Change in Serum Creatinine Levels
Description: Change in serum creatinine (Cr) levels after treatment with simvastatin
Time Frame: Baseline, 21 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Simvastatin, Dose Level 1 | Simvastatin, Dose Level 2 | Simvastatin, Dose Level 3
Number analyzed (Participants) | 16 | 12 | 2
mg/dL | 0.03 (0.03) | 0.04 (0.06) | -0.1 (0.1)

ADVERSE EVENTS:
Time Frame: 39 days
Description: Participants were assessed at day 0 (baseline), day 7, 14, 21 (treatment), day 25 (after taper)and day 39 (follow-up after discontinuation of treatment).
Groups:
- Simvastatin, Dose 1: Simvastatin given in a dose-escalating fashion to 3 sequential dosage groups (20 mg/day, 40 mg/day, 80 mg/day).
  Dose 1 = 20mg/day for 21 days, followed by 4-day drug taper.
- Simvastatin, Dose 2: Simvastatin given in a dose-escalating fashion to 3 sequential dosage groups (20 mg/day, 40 mg/day, 80 mg/day).
  Dose 2 = 40mg/day for 21 days, followed by a 4-day taper.
- Simvastatin, Dose 3: Simvastatin given in a dose-escalating fashion to 3 sequential dosage groups (20 mg/day, 40 mg/day, 80 mg/day).
  Dose 3 = 80mg/day for 21 days, followed by 4-day drug taper. Enrollment in this group discontinued early due to FDA warning re. high dose simvastatin
Arm/Group | Simvastatin, Dose 1 | Simvastatin, Dose 2 | Simvastatin, Dose 3
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/20 | 0/2
Other Adverse Events (participants affected / at risk) | 3/20 | 3/20 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin, Dose 1 (N=20) | Simvastatin, Dose 2 (N=20) | Simvastatin, Dose 3 (N=2)
sickle cell acute chest syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
sickle cell vaso-occlusive pain episode (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — vaso-occlusive pain event requiring hospitalization, parenteral opioid treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin, Dose 1 (N=20) | Simvastatin, Dose 2 (N=20) | Simvastatin, Dose 3 (N=2)
elevated serum creatine kinase level (General disorders) | 2 (2) | 3 (3) | 1 (1) — Increase in serum creatine kinase (CK) levels: 4 subjects: asymptomatic (AE, grade 1) 2 subjects: with myalgias (AE, grade 2)
sickle cell vaso-occlusive pain event (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) — vaso-occlusive pain event, requiring oral opioids, not hospitalized
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) — muscle pain associated with increase in serum creatine kinase level. occurred in 2 subjects: 1. simvastatin, 40mg/day, day 4: creatine kinase >2X UNL with muscle aches 2. simvastatin, 80mg/day, day 6: creatine kinase >4X UNL with muscle aches

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No